CLINICAL TRIAL: NCT04072679
Title: Evaluation of the Safety and Efficacy of Sintilimab Combined With IBI305 in the Treatment of Advanced Hepatocellular Carcinoma in a Single-center, One-arm, and Phase Ib Study
Brief Title: Safety and Efficacy Study of Sintilimab Combined With IBI305 in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI338B101
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Advanced Hepatocellular Carcinoma; Sintilimab; IBI305

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+IBI305 (Experimental): Sintilimab: 200mg (D1, q3w） IBI305: 7.5mg/kg or 15mg/kg (D1, q3w）
  Interventions: Drug: Sintilimab+IBI305

INTERVENTIONS:
Drug: Sintilimab+IBI305 — It includes dose escalation and dose expansion stage. 6-9 subjects will be enrolled in dose escalation stage for the safety and efficacy evaluation. Then select specific dose of IBI305 +Sintilimab 200mg/kg, expand to 36-39 patients for the further safety and efficacy study.The study treatment lasts up to 24 months.

SUMMARY:
This is a Phase Ib study to evaluate the safety, tolerability and efficacy of Sintilimab combined with IBI305 in patients with advanced hepatocellular carcinoma in China.

DETAILED DESCRIPTION:
This study is to evaluate the safety, tolerability and efficacy of Sintilimab combined with IBI305 in patients with advanced hepatocellular carcinoma in China.

Approximately 26-38 subjects with locally advanced or metastatic hepatocellular carcinoma will be enrolled in the study. It includes dose escalation and dose expansion stage. 12-18 subjects will be enrolled in dose escalation stage for the safety and efficacy evaluation. Then select specific dose of IBI305 +Sintilimab 200mg/kg, expand to 20 patients for the further safety and efficacy study.

The study treatment lasts up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Local advanced or metastatic hepatocellular carcinoma, confirmed by histology/cytology.
2. Barcelona Clinic Liver Cancer (BCLC) C. BCLC B, unsuitable for local treatments or local treatments failure.
3. Patients who failed to or unsuitable for the previously systemic chemotherapy, sorafenib, lenvatinib, regorafenib or similar drug failure (disease progression or toxicity intolerance).
4. At least one measurable lesion per RECIST V1.1 that has not been treated locally or that has progressed after local treatment.
5. Child-Pugh score ≤ 7 points.
6. ECOG：0 or 1.
7. Adequate organ and bone marrow function.

Exclusion Criteria:

1. With fibrous lamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma components in tumor tissues.
2. Have a history of hepatic encephalopathy or have a history of liver transplantation.
3. HBV DNA>2000 IU/ml or 104 copies/ml for acute or chronic active hepatitis B or hepatitis C; HCV RNA>103 copies/ml; both HbsAg and anti-HCV antibody are positive.
4. Esophageal or gastric varices bleeding caused by portal hypertension occurred in the past 6 months. Patients with endoscopy evidence of severe varices (G3) within 3 months. Patients with portal hypertension in high risk of bleeding evaluated by investigator.
5. History of venous thromboembolism in the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or any other history of severe thromboembolism. Implantable IV ports or catheter-derived thrombosis, superficial venous thrombosis, or thrombosis after conventional anticoagulant therapy are excluded. Prophylactic uses of low-dose aspirin or low molecular weight heparin is allowed.
6. Portal vein tumor thrombus (PVTT) involves both the main trunk and contralateral branch or upper mesenteric vein. Inferior vena cava tumor thrombus.
7. Uncontrolled high blood pressure, systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg after optimal medical treatment; Hypertensive crisis or history of hypertensive encephalopathy.
8. History of gastrointestinal perforation and/or fistula in the past 6 months, history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) , complicated by chronic diarrhea), Crohn's disease, ulcerative colitis or long-term chronic diarrhea.
9. History of interstitial pneumonia, drug-induced pneumonia, idiopathic pneumonia or active pneumonia. Allow radioactive pneumonia in the radiotherapy area.
10. Active tuberculosis (TB), who are receiving anti-tuberculosis treatment or who have received anti-tuberculosis treatment within 1 year before inclusion.
11. HIV infected (HIV 1/2 antibody positive).
12. Use of immunosuppressive drugs in the past 4 weeks, excluding the routes of topical glucocorticoids or physiological doses of systemic glucocorticoids (ie no more than 10 mg/day of prednisone or equivalent). Temporary use of glucocorticoids for dyspnea symptoms such as asthma and chronic obstructive pulmonary disease is allowed.
13. Have undergone major surgery (craniotomy, thoracotomy or open surgery) or unhealed wounds, ulcers or fractures within 4 weeks.
14. Previously received any anti-PD-1, anti-PD-L1/L2 antibodies, anti-CTLA4 antibodies, or other immunotherapy; previously received anti-VEGF monoclonal antibody treatment.
15. Female patients who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Incicende of Adverse Events (AEs) | 2 years
  Number of patients with AE, treatment-related AE (TRAE), immune-related AEs (irAE), AE of special interest (AESI), serious adverse event (SAE) assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Investigator assessed according to RECIST v1.1
Time to response (TTR) | 2 years
  Investigator assessed according to RECIST v1.1
Duration of response (DOR) | 2 years
  Investigator assessed according to RECIST v1.1
Disease control rate (DCR) | 2 years
  Investigator assessed according to RECIST v1.1
Progression free survival (PFS) | 2 years
  Investigator assessed according to RECIST v1.1
Overall Survival (OS) | 2 years
  Investigator assessed according to RECIST v1.1
Anti-drug antibody (ADA) | 2 years
  Immunogenicity measured by anti-drug antibody (ADA) for Sintilimab and IBI305

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou Zhou, Doctor, Principal Investigator — National Cancer Center/Cancer Hospital, China
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese ACademy of Medical Sciences and Peking Union Medical College, Beijing, China